CLINICAL TRIAL: NCT07391982
Title: Dose De-escalation in Prostate Radiotherapy Using an MR-Linac in 2 Fractions
Brief Title: Dose De-escalation in Prostate Radiotherapy Using an MR-Linac in Two Fractions
Acronym: DESTINATION 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: MRL Consortium (Unknown); Elekta Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M24DTI
Record Dates: First submitted 2025-10-02; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer (Adenocarcinoma)
Keywords: De-escalation; Radiotherapy; MR-Linac
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uniform dose SBRT (Other)
  Interventions: Radiation: uniform dose radiotherapy
- De-escalated dose SBRT (Other)
  Interventions: Radiation: De-escalated dose radiotherapy

INTERVENTIONS:
Radiation: uniform dose radiotherapy — 27 Gy dose in 2 fractions to the whole prostate+/- seminal vesicles with a 0mm PTV margin using MR-linac
  Arms: Uniform dose SBRT
Radiation: De-escalated dose radiotherapy — The benign prostate +/- SV CTV will receive 20 Gy in 2 fractions with a 0mm PTV margin using MR-linac. The intraprostatic tumor masses (on MRI) will receive 27 Gy in 2 fractions. A 4mm GTV to PTV margin will be added to the in-traprostatic MR visible tumour to form PTV 27Gy.
  Arms: De-escalated dose SBRT

SUMMARY:
The goal of this clinical trial is to find out whether lowering the radiation dose to parts of the prostate without visible tumor on MRI can reduce side effects while still effectively treating prostate cancer in men with low or intermediate-risk prostate cancer.

The main questions it aims to answer are:

* Does reducing the radiation dose to healthy prostate tissue lower the risk of bowel and urinary side effects?
* Can we maintain good cancer control by keeping a high dose for MRI-visible tumor areas?

Researchers will compare two treatment approaches:

* One group receives a uniform high dose to the entire prostate.
* The other group receives a lower dose to healthy prostate tissue and a high dose only to visible tumor areas.

Participants will:

* Receive two sessions of MRI-guided radiotherapy using an MR-Linac.
* Complete questionnaires about urinary, bowel, and sexual health before and after treatment.
* Have follow-up visits to monitor side effects and PSA levels for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged ≥18 years
2. Histological confirmation of prostate adenocarcinoma requiring radical radiotherapy
3. Gleason score 3+3, 3+4 or 4+3 (ISUP Grade groups (GG) 1, 2 or 3)
4. MRI-visible tumour(s) of PIRADS v2 grade 3 or higher and able to be delineated on T2 and diffusion-weighted imaging +/- dynamic contrast-enhanced imaging. Tumour nodule visible on MRI should be considered able to be boosted by treating clinician and <2.5cm in maximal dimension. MRI must be performed within 3 months of trial entry
5. The MRI-defined lesion must be confirmed as malignant on biopsies (any Gleason grade is sufficient as long as Gleason score is reported).
6. MRI stages mT1 and T2 or mT3a with ≤ 1mm tumour outside gland AND otherwise favourable intermediate risk characteristics (Gleason 3+3, 3+4)(as staged by AJCC TNM 2018)
7. PSA <20 ng/ml prior to starting androgen deprivation therapy (ADT).
8. WHO Performance status 0-2
9. Ability of the participant to understand and the willingness to sign a written informed consent (IC) form.
10. Ability/willingness to comply with the patient reported outcome questionnaires schedule throughout the study.

Exclusion Criteria:

1. Contraindications to MRI (e.g. pacemaker, potentially mobile metal implant, claustrophobia)
2. IPSS Score > 19
3. High grade disease (GG3) occult to MRI-defined lesion. As a guide, any pathology for which you would consider surveillance is allowed outside of the MRI-defined area.
4. Prostate volume >90cc
5. Comorbidities which predispose to significant toxicity (e.g. inflammatory bowel disease) or preclude long term follow up
6. Hip replacement, or other pelvic metalwork which causes artefact on diffusion-weighted imaging
7. Previous pelvic radiotherapy
8. Patients needing >6 months of ADT due to disease parameters.
9. Previous invasive malignancy within the last 2 years excluding basal or squamous cell carcinomas of the skin, low risk non-muscle invasive bladder cancer (assuming cystoscopic follow up now negative) or small renal masses on surveillance.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Acute GU toxicity | within 13 weeks of starting radiotherapy
  Physician-reported acute Grade 2 or higher CTCAE GU toxicity observed within 13 weeks of starting radiotherapy

SECONDARY OUTCOMES:
Dosimetry | During Radiotherapy treatment of 8 days
  Estimate the accumulated dose differences between treatment arms in terms of dose to prostate CTV, rectum, urethra and bladder
Late GI toxicity | 1 and 2 years after radiotherapy treatment
  Physician reported late GI toxicity according to CTCAE v5.0
Biochemical relapse-free survival | 2 years
  Assess biochemical relapse-free survival for 2 years
Severity of erectile dysfunction experienced by patient | Before radiotherapy treatment, and at 6, 12 and 24 months after radiotherapy treatment
  The IIEF-5 patient reported outcomes (PROs) assess the acute severity of erectile dysfunction
Acute GI toxicity | At baseline, after the last fraction, and 2, 4 and 12 weeks after radiotherapy treatment
  Physician reported acute GI toxicity according to CTCAE v5.0
Late GU toxicity | 1 and 2 years after radiotherapy treatment
  Physician reported late GU toxicity according to CTCAE v5.0
Late sexual toxicity | 1 and 2 years after radiotherapy treatment
  Physician reported late sexual toxicity according to CTCAE v5.0
Severity of urinary symptoms (GU) experienced by patient | Before radiotherapy treatment, after the last fraction, at 2, 4 and 12 weeks post-treatment, and at 6, 12 and 24 months after radiotherapy treatment
  The patient reported outcomes (PROs) International Prostate Symptoms Score (IPSS) assess the severity of urinary symptoms what the patient experiences
Health-related quality of life experienced by patient | Before start radiotherapy, week 4 and week 12, at 6, 12 and 24 months after radiotherapy treatment.
  The EPIC-26 patient reported outcomes (PROs) assess the health-related quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- The Netherlands Cancer Institute, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
It is intended that data will be shared within the MOMENTUM collaboration, between centres delivering treatment in the same way as DESTINATION2. Pseudonymised data will be stored within MOMENTUM for at least 5 years. Storage will be cloud based and as the treating centre we will have free access to the data and control over who else can assess it.
Time Frame: 5 years